CLINICAL TRIAL: NCT06783569
Title: A First-in-Human, Open-Label, Dose Escalation and Expansion Study of JR8603 in Patients With Advanced Solid Tumors
Brief Title: A First-in-Human Escalation and Expansion Study of Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: JiaRay Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JR8603-9101
Record Dates: First submitted 2025-01-07; First posted 2025-01-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors; Gastric Cancer; Esophagogastric Juction Cancer; Colorectal Cancer
Keywords: locally advanced solid tumors; metastatic solid tumors; intolerant to standard therapies; Mitomycin C
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1: Dose Escalation- will consist of accelerated titration followed by traditional 3+3 design. The accelerated titration portion may consist of up to 3 patients in the first 2 dose levels and the 3+3 ascending dose escalation portion will consist of 3 to 6 patients per dose level.
  Part 2: Dose Expansion- each cohort will be enrolled independently following a Simon's 2-Stage optimal design. In the first stage, 10 evaluable patients will be enrolled. If there is only 1 or no response in these 10 patients, the cohort will be stopped. Otherwise, 19 additional evaluable patients will be accrued to that cohort for a total of 29 evaluable patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Escalation Cohort - Dose Level -1 (Experimental): Dose Level -1: 1.7mg/m2. A Dose Level -1 cohort will be introduced if a dose reduction to a lower level is required.
  Interventions: Drug: JR8603
- Escalation Cohort - Dose Level 1 (Experimental): Dose Level 1: 3.3mg/m2.
  For Dose Levels 1 and 2, a single patient will be enrolled per dose level. If the patient in Dose Level 1 does not experience a Grade ≥2 adverse event (AE) that is not clearly attributed to an extraneous cause, such as the patient's underlying disease, other medical conditions, or concomitant medications or procedures during the dose-limiting toxicity (DLT) period, then Dose Level 2 will also be a single patient.
  If the patient in Dose Level 1 experiences a Grade ≥2 AE during the DLT period, then 2 additional patients will be added to Dose Level 1 and the remainder of the study will use 3+3 design rules.
  Interventions: Drug: JR8603
- Escalation Cohort - Dose Level 2 (Experimental): Dose Level 2: 7.0mg/m2. If Dose Level 2 is qualified to be a single patient, and the patient does not experience a Grade ≥2 AE during the DLT period, then Dose Level 3 will proceed and the study, thereafter, will utilize 3+3 design rules.
  If the patient in Dose Level 2 experiences a Grade ≥2 AE during the DLT period, then 2 additional patients will be enrolled in Dose Level 2 and evaluated using 3+3 design rules.
  Interventions: Drug: JR8603
- Escalation Cohort - Dose Level 3 (Experimental): Dose Level 3: 14.0mg/m2. From Dose Level 3 and thereafter, dose escalation will follow 3+3 design rules with 3 patients enrolled in each dose level. If 3 patients complete the DLT period with no DLTs, that dose level of JR8603 will be deemed safe, and another 3 patients will be treated at the next higher dose level.
  If 1 of the first 3 patients experiences a DLT, 3 more patients will be treated at the same dose level of JR8603.
  If 2 or more of the 3 to 6 patients in any dose level experience a DLT, dosing will stop at that level.
  Interventions: Drug: JR8603
- Escalation Cohort - Dose Level 4 (Experimental): Dose Level 4: 21.0mg/m2. Dose escalation will follow 3+3 design rules with 3 patients enrolled in each dose level. If 3 patients complete the DLT period with no DLTs, that dose level of JR8603 will be deemed safe, and another 3 patients will be treated at the next higher dose level.
  If 1 of the first 3 patients experiences a DLT, 3 more patients will be treated at the same dose level of JR8603.
  If 2 or more of the 3 to 6 patients in any dose level experience a DLT, dosing will stop at that level.
  Interventions: Drug: JR8603
- Escalation Cohort - Dose Level 5 (Experimental): Dose Level 5: 28.0mg/m2. Dose escalation will follow 3+3 design rules with 3 patients enrolled in each dose level. If 3 patients complete the DLT period with no DLTs, that dose level of JR8603 will be deemed safe, and another 3 patients will be treated at the next higher dose level.
  If 1 of the first 3 patients experiences a DLT, 3 more patients will be treated at the same dose level of JR8603.
  If 2 or more of the 3 to 6 patients in any dose level experience a DLT, dosing will stop at that level.
  Interventions: Drug: JR8603
- Escalation Cohort - Dose Level 6 (Experimental): Dose Level 6: 35.0mg/m2. Dose escalation will follow 3+3 design rules with 3 patients enrolled in each dose level.
  If 1 of the first 3 patients experiences a DLT, 3 more patients will be treated at the same dose level of JR8603.
  If 2 or more of the 3 to 6 patients in any dose level experience a DLT, dosing will stop at that level.
  Interventions: Drug: JR8603
- Expansion Cohort 1 (Experimental)
  Interventions: Drug: JR8603
- Expansion Cohort 2 (Experimental)
  Interventions: Drug: JR8603

INTERVENTIONS:
Drug: JR8603 — IV infusion on Days 1, 8, and 15 of continuous 28-day cycles

SUMMARY:
The goal of this clinical trial is to learn if the investigational drug (JR8603) is safe and effective in treating patients with solid tumors after their initial rounds of treatment with other drugs did not work.

DETAILED DESCRIPTION:
This is a 2-part, first-in-human, open-label study to determine the safety and tolerability and preliminary efficacy of JR8603 in patients with locally advanced or metastatic solid tumors who have progressed after or are intolerant to standard therapies. The study will include a Dose Escalation Part and a Dose Expansion Part. JR8603 will be administered as a short IV infusion on Days 1, 8, and 15 of continuous 28-day cycles. Safety and tolerability of JR8603 will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. All patients will be assessed for response using Response Criteria for Evaluation in Solid Tumors (RECIST) v1.1, with computed tomography (CT) or magnetic resonance imaging (MRI) occurring at screening within 28 days of first dose, then every 8 weeks (±7 days) after Cycle 1 Day 1 (C1D1) for the first year and every 12 weeks (±7 days) thereafter. Serial blood samples for determination of PK will be collected.

ELIGIBILITY:
Inclusion Criteria

Patients who meet ALL the following inclusion criteria will be eligible to participate in the study:

1. ≥18 years of age.
2. Histologically confirmed, locally advanced, or metastatic solid tumor which has progressed on, or patients intolerant to, all standard therapy, or no standard therapy available, or it is documented that the therapy is refused by the patient.
3. Measurable disease per RECIST v1.1.
4. Life expectancy ≥3 months.
5. Adequate organ and bone marrow function defined by:

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L (≥1500/mm3)
   2. Platelet count ≥100 × 109/L (≥100,000/mm3) (no platelet transfusion within 14 days prior to enrollment)
   3. Total bilirubin ≤1.5 × upper limit of normal (ULN), unless known Gilbert syndrome (≤3 × ULN) has been diagnosed
   4. AST and ALT ≤2.5 × ULN or ≤5 × ULN for patients with known liver metastases
   5. Estimated creatinine clearance by the Cockcroft-Gault or estimated glomerular filtration rate (eGFR) of ≥60 mL/min
   6. International Normalized Ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤1.5 × ULN. If a patient is receiving anticoagulant therapy, PT and aPTT must be within therapeutic range of intended use of anticoagulants
6. Patients with treated, stable central nervous system (CNS) metastases (including leptomeningeal carcinomatosis) are allowed if there is no evidence of progression for at least 4 weeks after CNS-directed treatment as ascertained by clinical examination and brain imaging.
7. Resolution of any clinically significant toxic effects of prior therapy to Grade ≤1 according to the NCI CTCAE v5.0 (exception of alopecia and Grade 2 peripheral neuropathy).
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Willingness of men and women of reproductive potential to observe conventional and effective birth control methods with failure rates of <1% for the duration of treatment and for at least 6 months for women and at least 3 months for men following the last dose of study treatment (this must include a barrier method such as condom or diaphragm with spermicidal gel). Women of reproductive potential are defined as following menarche and who are not postmenopausal (and 2 years of nontherapy-induced amenorrhea or surgically sterile). For male patients with a nonpregnant female partner of childbearing potential and a woman of childbearing potential, 1 of the following highly effective birth control methods with a failure rate of less than 1% per year when used consistently and correctly are recommended:

   1. Combined estrogen and progestin containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or transdermally
   2. Progestin-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant
   3. Intrauterine device
   4. Intrauterine hormone-releasing system
   5. Bilateral tubal occlusion/ligation
   6. Vasectomized partner
   7. Sexual abstinence Note: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient. Birth control methods unacceptable for this study include the following:

   <!-- -->

   1. Periodic abstinence (calendar, symptothermal, or post-ovulation methods)
   2. Withdrawal (coitus interruptus)
   3. Spermicide only
   4. Lactational amenorrhea method Egg and sperm donation or banking is prohibited during the duration of participation on this protocol and for 90 days after the last dose of study drug. 10. A negative serum pregnancy test at screening and a negative (serum or urine) pregnancy test within 72 hours before the first dose of study drug (female patients of childbearing potential only). If the urine test is positive or cannot be confirmed negative, a serum pregnancy test will be required and must be negative for the patient to be eligible.

11. Willing and able to provide informed consent and comply with protocol requirements for the duration of the study.

Specific Inclusion Criteria for Expansion Cohorts:

To be eligible during the dose expansion part of the study, patients must meet 1 of the following 2 criteria:

Expansion Cohort 1: Documented locally advanced or metastatic gastric or

EGJ cancer which has progressed on or after standard therapy or patient is intolerant to standard therapy or patient refuses therapy. Standard therapy options are described in (Wang,2024):

* Prior systemic standard therapy for patients with HER2-positive gastric or EGJ cancer should include trastuzumab plus chemotherapy (fluorouracil plus platinum), mono-chemotherapy (eg., paclitaxel, docetaxel, irinotecan), and other monotherapy (eg., VEGF targeted agents, anti-PD-1 or PD-L1).
* Prior system standard therapy for patients with HER2-negative gastric or EGJ cancer should include fluorouracil plus platinum or in combination with anti-PD-1, mono-chemotherapy (eg., paclitaxel, docetaxel, irinotecan) and VEGF targeted therapy.

Expansion Cohort 2: Documented locally advanced or metastatic colorectal cancer which has progressed on or after standard therapy or patient is intolerant to standard therapy, or patient refuses therapy. Standard treatment options are described in (Association NHCOTPROCSOOCM,2023):

* Prior systemic standard therapy for patients with MMR-deficient (dMMR)/microsatellite instability-high (MSI-H): pembrolizumab for 1st line therapy, no standard therapy for 2nd and 3rd line therapy.
* Prior system standard therapy for patients with microsatellite stability (MSS) or microsatellite instability-low (MSI-L)/proficient mismatch repair (pMMR), RAS and BRAF wild-type (WT) should include cetuximab or bevacizumab monotherapy or in combination with FOLFOX/FOLFIRI/CAPEOX, and monotherapy (eg., regorafenib, fruquintinib, trifluridine tipiracil).
* Prior system standard therapy for patients with MSS or MSI-L/pMMR, RAS and BRAF mutation: should include bevacizumab monotherapy or in combination with FOLFIRI, and monotherapy (eg., regorafenib, fruquintinib, trifluridine tipiracil).

Exclusion Criteria Patients who meet any of the following exclusion criteria will be excluded from participation in the study:

1. Any condition that in the opinion of the Investigator would place the patient at an unacceptable risk or cause the patient to be unlikely to fully participate or comply with study procedures.
2. Received systemic anticancer chemotherapy, targeted agents, antibody therapy for cancer, immunotherapy for cancer, hormonal therapy, or an investigational agent within 2 weeks or 5 half-lives (whichever is shorter) prior to start of study drug treatment.
3. Major surgery within 3 weeks prior to start of study drug treatment.
4. Radiation therapy within 4 weeks prior to start of study drug treatment (palliative radiation or stereotactic radiosurgery within 7 days prior to start of study drug treatment). Patients must have recovered from all acute radiotherapy-related toxicities.
5. Severe or unstable cardiac conditions including, but not limited to, congestive heart failure (New York Heart Association Class III or IV), ischemic heart disease, uncontrolled hypertension, uncontrolled cardiac arrhythmia requiring medication (Grade ≥2, according to NCI CTCAE v5.0), myocardial infarction within 6 months prior to starting study drug treatment, congenital long QT syndrome or QT interval corrected for heart rate using Fridericia's formula (QTcF) >470 msec at screening, and any other significant or unstable concurrent cardiac illness.
6. Severe or unstable medical condition including uncontrolled diabetes or unstable psychiatric condition.
7. Has a history of another active malignancy (a second cancer) within the previous 2 years except for localized cancers that are not related to the current cancer being treated, are considered cured, and, in the opinion of the Investigator, present a low risk of recurrence. These exceptions include, but are not limited to, basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
8. Active infection requiring systemic therapy (including asymptomatic infections with positive virus titers and the Investigator's judgment that worsening of the condition is likely with study drug or the condition will impair or prohibit a patient's participation in the study).
9. Known human immunodeficiency virus, hepatitis B virus (HBV) (i.e., hepatitis B surface antigen positive), or hepatitis C virus (HCV) (i.e., detectable HCV ribonucleic acid [RNA]). Note: Patients with a prior history of treated HBV infection who are antigen negative, patients with a prior history of treated HCV infection who are HCV RNA undetectable, or patients with HIV who are on stable anti-retroviral therapy and have an undetectable viral load may be enrolled.
10. Pregnant (or intending to become pregnant) or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (Including Serious Adverse Events) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  The severity of all AEs will be graded according to the NCI CTCAE v5.0 criteria.
Dose-Limiting Toxicity (DLT) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Incidence of DLTs
Maximum tolerated dose (MTD) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Evaluated based on DLT-Evaluable patients in part 1 Dose Escalation
Dose Expansion - to assess preliminary evidence of efficacy for each cohort | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Measured by Overall Response Rate (ORR) as defined by RECIST v1.1.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Defined as the proportion of patients with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) per RECIST v1.1
Assess Plasma concentrations and relevant PK parameters for JR8603 and the active metabolite (mitomycin C) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Will be assessed based on blood samples collected from patients during the study.
Time to Response (TTR) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Defined as the time from the date of the first dose to the date at which criteria are first met for Complete Response (CR) or Partial Response (PR) per RECIST v1.1.
Duration of Response (DOR) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Defined as the time from the start of the first response (CR or PR) to the first occurrence of progressive disease per RECIST v1.1 or death due to any cause
Disease Control Rate (DCR) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Defined as the proportion of patients whose best overall response is a CR, PR, or stable disease (SD)
Progression-free survival (PFS) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Defined as the time from the first dose of JR8603 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | From study drug administration until 28 (±7) days after the last dose of study drug, up to approximately 1 year
  Defined as the time from the date of the first dose of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical University Cancer Hospital, Harbin, Heiljiang Province
  - Liaoning Cancer Hospital, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided